CLINICAL TRIAL: NCT00526123
Title: A Randomized, Open-label Comparison of the Performance and Longevity of a Split-tip Versus a Symmetric Tip Hemodialysis
Brief Title: Dialysis Catheter Comparative Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tyco Healthcare Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 341.26
Record Dates: First submitted 2007-09-05; First posted 2007-09-06 (Estimated); Results first posted 2013-01-07 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: End Stage Renal Disease
Keywords: Dialysis; Dialysis Catheter; Kidney Disease; Dialysis Clinic; Chronic Catheter; Catheter; Kidney
MeSH Terms: conditions — Kidney Failure, Chronic; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): symmetric tip catheter
  Interventions: Device: Symmetric Tip Catheter
- 2 (Active Comparator): conventional split-tip catheter
  Interventions: Device: Conventional Split-tip Catheter

INTERVENTIONS:
Device: Symmetric Tip Catheter — Dialysis catheter
  Arms: 1
Device: Conventional Split-tip Catheter — Dialysis Catheter
  Arms: 2

SUMMARY:
The purpose of this clinical trial is to compare the longevity of two dialysis catheters.

DETAILED DESCRIPTION:
This study is a multi-center, randomized, prospective, open-label, clinical study comparing a conventional split-tip catheter and a symmetric tip catheter in subjects undergoing hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older.
* Subject must meet labeled indication for hemodialysis.
* Subject must have End Stage Renal Disease (ESRD).
* Subject must have a patent right or left internal jugular vein.
* Subject treatment plan must require chronic hemodialysis treatments 3 times per week for a minimum of 6 weeks.
* Subject must give written informed consent.

Exclusion Criteria:

* Subjects who are concurrently enrolled in any Randomized Clinical Trial (RCT) or those that may enroll in a RCT during the course of the study, or subjects who have been previously randomized into this clinical study.
* Subjects with active infection at the time of study enrollment.
* Subjects with a known sensitivity to heparin, or previous incidence of heparin-induced thrombocytopenia.
* Subjects with uncontrolled abnormal coagulation parameters and are at additional risk for clotting or excessive bleeding.
* Subjects who are known or suspected to be pregnant at the time of study enrollment or plan to get pregnant during the study period.
* Subjects for whom performing dialysis at flow rates up to 450 mL/min would be contraindicated for any reason.
* Subject unable or unwilling to commit to follow-up visits and study procedures throughout the course of the study.
* Subjects who, in the opinion of the Investigators, are not appropriate candidates for the study based upon current or past medical history, or negative past experience with either of the study catheters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2007-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klemens B Meyer, MD, Principal Investigator
Locations (14):
- United States (14):
  - Nephrology Associates, P.C., Birmingham, Alabama
  - Southwest Kidney Institute, Phoenix, Arizona
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - SUNY Stony Brook Medical Center, Stony Brook, New York
  - Eastern Nephrology Associates, Greenville, North Carolina
  - Eastern Nephrology Associates, New Bern, North Carolina
  - Boice-Willis Clinic, Rocky Mount, North Carolina
  - Dialysis Access Group of Wake Forest University, LLC, Winston-Salem, North Carolina
  - Toledo Hospital, Toledo, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Nephrology Associates - Lankenau Hospital, Wynnewood, Pennsylvania
  - Columbia Nephrology Associates, Columbia, South Carolina
  - Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with ESRD requiring hemodialysis via a chronic hemodialysis catheter at least 3x weekly for a minimum of 6 weeks were recruited from the clinical study sites. Participating sites included hospitals and private medical clinics. Subjects were enrolled from September 2007 through January 2011
Pre-assignment Details: Patients that met all of the eligibility criteria were enrolled and were randomized 1:1 to either the symmetric tip or split-tip catheter group. Enrolled subjects were further stratified via subject ID by new catheter insertion versus catheter exchange.
Groups:
- Symmetric Tip: symmetric tip hemodialysis catheter
- Split-tip: split-tip hemodialysis catheter
Period: Overall Study
Arm/Group | Symmetric Tip | Split-tip
Started | 303 (Intent-to-Treat population) | 296 (Intent-to-Treat population)
Completed | 39 | 50
Not Completed | 264 | 246

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symmetric Tip | Split-tip | Total
Number analyzed (Participants) | 303 | 296 | 599
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 189 | 180 | 369
  >=65 years | 114 | 115 | 229
Age Continuous [Mean (Standard Deviation); unit: years] | 60.0 (14.49) | 58.9 (15.34) | 59.5 (14.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 149 | 309
  Male | 143 | 147 | 290
Region of Enrollment [Number; unit: participants]
  United States | 303 | 296 | 599

OUTCOME MEASURES:

1. Primary Outcome: First Catheter Induced Complication
Description: % of participants that did not experience a catheter induced complication at the specified Outcome Measure Time Frame.
Time Frame: 30 days
Population: Number of participants is derived from the 'per protocol' population defined as those subjects that were randomized and have at least one post baseline measurement for the primary efficacy endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Symmetric Tip | Split-tip
Number analyzed (Participants) | 285 | 283
percentage of participants | 78 | 77

2. Secondary Outcome: Inadequate Flow Rates Requiring Surgical/Radiological Intervention
Description: Number of events per study group in which the first catheter induced complication was 'inadequate flow requiring surgical/radiological intervention'.
Time Frame: 35 weeks
Population: Number of participants is derived from the 'intent to treat' population defined as those subjects that were randomized.
Measure: Number; unit: events
Arm/Group | Symmetric Tip | Split-tip
Number analyzed (Participants) | 303 | 296
events | 18 | 29

3. Primary Outcome: First Catheter Induced Complication
Description: % of participants that did not experience a catheter induced complication at the specified Outcome Measure Time Frame.
Time Frame: 60 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Symmetric Tip | Split-tip
Number analyzed (Participants) | 285 | 283
percentage of participants | 66 | 69

4. Primary Outcome: First Catheter Induced Complication
Description: % of participants that did not experience a catheter induced complication at the specified Outcome Measure Time Frame.
Time Frame: 245 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Symmetric Tip | Split-tip
Number analyzed (Participants) | 285 | 283
percentage of participants | 40 | 48

5. Secondary Outcome: Average Number of Line Reversals Per Subject
Description: Average number of times the dialysis lines were reversed per subject to deliver dialysis treatments
Time Frame: 35 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Symmetric Tip | Split-tip
Number analyzed (Participants) | 285 | 283
events | 6.5 (18.87) | 8.0 (21.01)

6. Secondary Outcome: Frequency of Clinician Interventions for Catheter Malfunction and Infection
Description: Average number of times clinician intervention was required for either catheter malfunction or infection
Time Frame: 35 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Symmetric Tip | Split-tip
Number analyzed (Participants) | 285 | 283
events | 8.2 (12.22) | 10.0 (15.89)

7. Secondary Outcome: Primary Failure Rate
Description: The percentage of catheters unable to deliver adequate blood flow of at least 300 mL/min for at least 50% of measurements during the first attempted dialysis session.
Time Frame: First dialysis session with study catheter
Population: Number of participants was derived from the 'per protocol' population defined as those subjects that were randomized, had a study catheter inserted, and have at least one post baseline measurement for the primary efficacy endpoint.
Measure: Number; unit: percentage of catheters
Arm/Group | Symmetric Tip | Split-tip
Number analyzed (Participants) | 285 | 283
percentage of catheters | 3.9 | 4.9

8. Secondary Outcome: Reliability of the Catheter
Description: Percentage of study visits in which the median blood flow rate was greater than or equal to 300 mL/min.
Time Frame: 35 Weeks
Population: Number of participants was derived from the 'per protocol' population defined as those subjects that were randomized, had the study catheter inserted, and have at least one post baseline measurement for the primary efficacy endpoint.
Measure: Mean (Standard Deviation); unit: percentage of study visits
Arm/Group | Symmetric Tip | Split-tip
Number analyzed (Participants) | 285 | 283
percentage of study visits | 90.6 (20.10) | 86.9 (23.37)

ADVERSE EVENTS:
Time Frame: Immediately following study catheter insertion any adverse effect that was determined by the Investigator to be possibly or probably related to the study catheter or study procedures was collected.
Arm/Group | Symmetric Tip | Split-tip
Serious Adverse Events (participants affected / at risk) | 11/303 | 4/296
Other Adverse Events (participants affected / at risk) | 0/303 | 0/296
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Symmetric Tip (N=303) | Split-tip (N=296)
Bacteremia (Infections and infestations) | 1 (2) | 0 (0)
Catheter Infection (Infections and infestations) | 2 (2) | 0 (0)
Catheter-related bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Catheter-related blood stream infection (CRBSI) (Infections and infestations) | 1 (1) | 0 (0)
Exit site infection (Infections and infestations) | 1 (1) | 0 (0)
Fever of unknown origin, bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Gram negative bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infection, permcath associated bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Methicillin resistant staphylococcus aureus-sepsis (MRSA) (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary embolism (PE) (Vascular disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (3)
Staph aureus bacteremia (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
SPONSOR shall have the right to review and comment on such publication with respect to disclosure of SPONSOR Confidential Information prior to submission and review, and no such SPONSOR Confidential Information shall be disclosed therein without SPONSOR's express written consent. Such review and comment will be provided within 30 calendar days from the date of receipt by the SPONSOR. Investigator shall delete any SPONSOR confidential information contained in such publication.